CLINICAL TRIAL: NCT02591121
Title: Clinical Evaluation To Determine The Expected Values Distribution Of Procalcitonin For The RAMP® Procalcitonin Test In A Healthy Reference Population (PRO-H)
Brief Title: Procalcitonin Test Reference Range Determination
Acronym: PRO-H
Status: Completed | Type: Observational
Sponsor: Response Biomedical Corp. (Industry)
Responsible Party: Sponsor
Other Study IDs: CSP025
Record Dates: First submitted 2015-10-23; First posted 2015-10-29 (Estimated); Last update posted 2015-11-16 (Estimated); Status verified 2015-10

CONDITIONS: Healthy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No

SUMMARY:
Prospective, single-centre study in healthy volunteers to establish a reference range for the RAMP Procalcitonin (PCT) test. The primary objective of this study is to establish the reference range for measurement of PCT levels using the RAMP Procalcitonin test.

DETAILED DESCRIPTION:
Healthy volunteers who meet eligibility criteria and have provided informed consent will be enrolled in this study. Each participant will be required to donate 1 blood sample via standard venipuncture into an EDTA (lavender top) tube for testing on one occasion. The maximum trial duration for each participant is one visit/occasion. Sample collection will take place within a single clinical session. The maximum trial duration for each participant is one clinic session.

ELIGIBILITY:
Inclusion Criteria:

* Apparently healthy (as determined by a subject questionnaire) males or females, of any race
* >18 years of age
* Willing to voluntarily agree to sign a consent form

Exclusion Criteria:

* Meets the definition for one or more of Systematic Inflammatory Response Syndrome (SIRS), Sepsis, Severe Sepsis, Septic Shock and/or Multiple Organ Dysfunction Syndrome (MODS) as defined by The American College of Chest Physicians (ACCP) and the Society of Critical Care Medicine (SCCM) consensus conference in 1992.
* Current diagnosis, or history, of any underlying major medical condition such as heart disease, hypertension/hypotension, stroke, renal disease, chronic obstructive pulmonary disorder, diabetes, bleeding disorders, hypercalcitoninemia, HIV, etc.
* Bacterial, fungal or malaria infection within previous 12 months
* Have experienced or undergone trauma, surgery, cardiac shock and/or a burn within previous 3 months
* Current diagnosis of cancer and/or has undergone Immunotherapy which stimulates cytokines in the previous 12 months
* Hospitalization (for >24 hours) within previous 3 months
* Currently pregnant or nursing a child
* Unable, or unwilling, to provide required blood sample for testing
* Non-compliance to the protocol or inclusion criteria
* Investigator believes subject is unsuitable for inclusion in the trial (i.e. has major condition(s) or other reason(s) that could limit their ability to participate in the study; or impact the scientific integrity of the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy normal
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2015-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Procalcitonin value for healthy reference subjects | Subjects will be followed for duration of one blood draw from one visit only; study enrollment will occur over 21 days.
  Procalcitonin value for each subject will be determined within 2 hours of phlebotomy. At study completion all data obtained will be compiled and a 95th percentile value determined.

CONTACTS AND LOCATIONS:
Overall Officials: Azar Azad, Principal Investigator — Mount Sinai Services
Locations (1):
- Mt. Sinai Hospital, Toronto, Ontario, Canada